CLINICAL TRIAL: NCT06583577
Title: 3D Ostomy Simulation for Patient Education
Brief Title: Ostomy Simulation for Patient Education Prior to Urologic Bowel Diversion Surgeries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Device Feasibility
Other Study IDs: 00020255
Record Dates: First submitted 2024-08-01; First posted 2024-09-04 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Ostomy; Ileal Conduit
Keywords: Patient education; Simulation; Quality of life; Ostomy adjustment

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to two treatment groups. The experimental group will receive preoperative hands on education on stoma care using a new 3D model. The comparator group will receive standard preoperative education.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The post-operative soma care nurses and statistician will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D model simulator preoperative education (Experimental): Participants will receive standard preoperative education regarding ostomy care enhanced by the hands on use of a the ostomy simulator.
  Interventions: Device: 3D Ostomy simulator
- Standard preoperative education (No Intervention): Participants will receive standard preoperative education.

INTERVENTIONS:
Device: 3D Ostomy simulator — The ostomy simulator is 3D printed model created in collaboration with Earl E. Bakken Medical Devices Center at the University of Minnesota. The anatomically accurate model is created by analyzing de-identified segmental imaging after bowel diversion surgeries. The Stratasys J750 Polyjet 3D Printer is utilized to create the simulator using usual synthetic material.
  Arms: 3D model simulator preoperative education

SUMMARY:
The purpose of this study is to evaluate the feasibility of using a realistic and anatomically accurate 3D printed simulation model for urologic bowel diversion patient education. Using a randomized two group design, we aim to determine whether the use of this model enhances patient knowledge, self-care skills, and confidence in ostomy care. We will also evaluate changes in quality of life (QOL) and patient satisfaction comparing patients exposed to the 3D model to those receiving standard of care.

The secondary aim of the study is to examine the differences between groups on patient outcomes including hospital duration, mortality, emergency/urgent health care visits, readmissions, and infections.

Participants will be educated using 3D model simulation as part of their preoperative education (experimental group) or have standard education without using the simulation model (comparator group). Both groups will complete quality of life (QOL), ostomy adjustment, and satisfaction with education surveys during their preoperative education visit and again during their routine follow-up visits (a) within 3 weeks after surgery, (b) between 5- 8 weeks after surgery, and (c) at approximately 3 months after surgery.

DETAILED DESCRIPTION:
Inclusion Criteria:

Age>18 and planning to undergo bowel diversion urologic surgery.

Exclusion Criteria: Current or prior ostomy formation, cognitive function causing inability to care for stoma, current pregnancy.

Radom allocation and concealment: During a regularly schedule preoperative clinic visit participants that consent to the study will be asked to complete a short 36 item quality-of-life questionnaire (SF-36). The participant then be placed in either the experimental or comparator group using a random method similar to flipping a coin. Random allocation sequencing will be predetermined by a database specialist, who has no other role in the study. Therefore, all study staff, clinic staff and investigators will be blinded to the allocation sequencing, and will not be able to influence the group participants are assigned to.

Preoperative education: The clinic staff will provide participants with preoperative education according to their group assignment. Participants in the experimental group, will receive standard ostomy education supplemented by use of the simulation model. Those allocated to the comparator group will receive standard preoperative education.

Surveys: During the preoperative visit prior to receiving education, all participants will be asked to complete a quality of life survey, the SF-36. After the education, participants will be asked to complete the Ostomy Adjustment scale (OAS), and a visual analog scale (VAS) indicating their satisfaction with the ostomy education.

During regular postoperative visits within 3 weeks, between 5-8 weeks and approximately 3 months after leaving the hospital, participants will be asked to complete the SF-36, the OAS, and VAS. All study procedures will be conducted at the surgeon's clinic.

ELIGIBILITY:
Inclusion Criteria:

* Age>18, undergoing bowel diversion urologic surgery.

Exclusion Criteria:

* Current or prior ostomy formation, cognitive function causing inability to care for stoma, current pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Develop 3D printed model for urologic bowel diversion | Models were created and approved prior to start of the project
  3D printed model for urinary bowel diversion education
Quality of life using SF-36 scale | Preoperatively before education and within 3 weeks post hospital discharge, 5-8 weeks post hospital discharge, approximately 3 months post hospital discharge.
  Determine differences between groups in QOL using the (36-Item Short Form Health Survey)SF-36 Scale.
Adjustment of Ostomy | Preoperatively after education and within 3 weeks post hospital discharge, 5-8 weeks post hospital discharge, approximately 3 months post hospital discharge.
  Determine differences between groups in adjustment to ostomy using the ostomy adjustment scale (OAS) Scale.
Satisfaction with ostomy education | Preoperatively after education and within 3 weeks post hospital discharge, 5-8 weeks post hospital discharge, approximately 3 months post hospital discharge.
  Determine differences between groups in adjustment to ostomy using the Visual Analog Scale VAS Scale.

SECONDARY OUTCOMES:
Post operative hospital duration | Day the patient is deemed ready for hospital discharge, up to 52 weeks
  Number of postoperative days until participant is deemed ready for hospital discharge
In-hospital mortality | Up to 12 weeks
  Participant dies prior to discharge from hospital
Unplanned visit to urgent healthcare after discharge from the hospital | Measured at 3 weeks and 3 months
  Participant goes to urgent care, emergency room
Hospital readmission after discharge from the hospital. | Measured at 3 weeks and 3 months
  Patient has hospital admission due to ostomy surgery
Surgical site infection | Measured at 3 weeks and 3 months
  Diagnosis of surgical site infection requiring treatment

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No